CLINICAL TRIAL: NCT03137199
Title: A Phase I, Trial to Evaluate the Safety, Tolerability, and Potential Efficacy of Allogeneic Human Mesenchymal Stem Cell Infusion in Patients With Mild Asthma
Brief Title: Allogeneic Human Cells (hMSC) Via Intravenous Delivery in Patients With Mild Asthma
Acronym: ASTEC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: First cohort completed. Per sponsor decision.
Sponsor: Marilyn Glassberg (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Sponsor-Investigator, Marilyn Glassberg, Professor of Medicine, Surgery, and Pediatrics, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20160350
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Asthma
Keywords: stem cell; mesenchymal stem cell; lung; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: a first group of 3 patients will receive a lower dose of 20 million hMSCs, followed by a second group of 3 patients to receive a dose of 100 million hMSCs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group receiving 20 million hMSCs (Experimental): 3 patients will receive a single administration of allogeneic hMSCs: 20 x106 (20 million) cells delivered via peripheral intravenous infusion
  Interventions: Biological: hMSCs
- Group receiving 100 million hMSCs (Experimental): 3 patients will receive a single administration of allogeneic hMSCs: 1 x108 (100 million) cells delivered via peripheral intravenous infusion
  Interventions: Biological: hMSCs

INTERVENTIONS:
Biological: hMSCs — intravenous infusion of bone marrow-derived allogeneic stem cells
  Other Names: allogeneic mesenchymal stem cell

SUMMARY:
A Phase 1 investigation will be performed to test the safety of two doses of bone marrow-derived MSCs (20,000,000 and 100,000,000) administered via peripheral intravenous infusion.

DETAILED DESCRIPTION:
A Phase 1 investigation will be performed to test the safety of two doses of bone marrow-derived MSCs (20,000,000 and 100,000,000) administered via peripheralintravenous infusion.

Group 1: 3 subjects will receive a single administration of allogeneic hMSCs: 20 million cells delivered via peripheral intravenous infusion Group 2: 3 subjects will receive a single administration of allogeneic hMSCs: 100 million cells delivered via peripheral intravenous infusion Interim safety analysis will be performed four weeks after the 1st subject is enrolled in each cohort. Continued safety and tolerability with review of adverse events (AEs) will be assessed at each visit. Efficacy parameters (pulmonary function tests, diffusing capacity (DLCO), lung volumes, 6-minute walk test (6MWT), and dyspnea/quality of life [QOL] questionnaires) will be assessed every 12 weeks until study completion. Clinical laboratory tests to assess safety will be performed at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* be between 18 and 65 years at the time of signing the Informed Consent
* have a clinical diagnosis of asthma prior to screening in accordance with the guidelines of the American Thoracic Society/European Respiratory Society
* ACQ over 1.25
* have a smoking history of less than 10 pack-years total and have not been smoking for at least the last 12 months
* Perform a positive methacholine challenge at screening and repeat positive methacholine challenge at baseline visit (14 days later)
* Have normal or mild obstructive spirometry
* Have normal right heart function as documented by Doppler echo or right heart catheterization
* If female, be surgically sterile, post-menopausal (more than 1 year), or practice double barrier methods of birth control
* Subjects may receive non-drug therapies including oxygen supplementation no greater than 2L/minute, and pulmonary rehabilitation
* Subjects may be on standard of care asthma medications including inhaled corticosteroids-long acting beta agonist at a dose not greater than 1 mg of a fluticasone equivalent

Exclusion Criteria:

* Have any active infection that is not treated
* Be unable to perform any of the assessments required for endpoint analysis.
* currently receive (or have received within four weeks of screening) experimental agents for the treatment of asthma
* be actively listed (or expecting to be listed in the near future) for transplant of any organ
* Have clinically important abnormal screening laboratory values : blood screening tests (Hematology, Chemistry, CBC including Eosinophil count) results that are not within normal limits (according to UMHC Laboratory Reference Ranges) Have a serious comorbid illness that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study
* Have known allergies to penicillin or streptomycin
* Be an organ transplant recipient
* Have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma
* Have a non-pulmonary condition that limits lifespan to less than a year.
* Have a history of drug or alcohol abuse within the past 24 months.
* Be serum positive for HIV, hepatitis BsAg or Viremia hepatitis C
* Be currently participating (or have participated within the previous 30 days) in an investigational therapeutic or device trial.
* Have hypersensitivity to dimethyl sulfoxide (DMSO)
* Have a resting oxygen saturation (SpO2) on room air of more than 93% at sea level or more than 88% at an altitude above 5,000 feet above sea level (1524 meters)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Number of Participant with treatment emergent serious adverse events | Week 4 post infusion
  as defined as the incidence of any treatment-emergent serious adverse events; these are a composite of death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities

SECONDARY OUTCOMES:
Difference in lung function | Participants will be followed from 1 week to an expected average of 48 weeks following infusion
  Difference in FEV1 Variability in morning peak expiratory flow measurements
  Difference in frequency of acute exacerbations defined as:
  hospitalizations, missed work days, and/or oral steroids for more than 3 days Decrease in fractional excretion of inhaled NO (FENO; less than 50 ppb)
Decrease in peripheral eosinophilia | Participants will be followed from 1 week to an expected average of 48 weeks following infusion
  Decrease in number of peripheral eosinophils
Difference in subject reported dyspnea and quality of life assessments | Participants will be followed from 1 week to an expected average of 48 weeks following infusion
  Difference in subject reported dyspnea and quality of life assessments:
  Asthma Control Test (ACT) and Asthma Control Questionnaire (ACQ)
Death from any cause | Participants will be followed from 1 week to an expected average of 48 weeks following infusion
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn K Glassberg, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szefler SJ, Wenzel S, Brown R, Erzurum SC, Fahy JV, Hamilton RG, Hunt JF, Kita H, Liu AH, Panettieri RA Jr, Schleimer RP, Minnicozzi M. Asthma outcomes: biomarkers. J Allergy Clin Immunol. 2012 Mar;129(3 Suppl):S9-23. doi: 10.1016/j.jaci.2011.12.979. PMID 22386512
- [Background] Malmstrom K, Rodriguez-Gomez G, Guerra J, Villaran C, Pineiro A, Wei LX, Seidenberg BC, Reiss TF. Oral montelukast, inhaled beclomethasone, and placebo for chronic asthma. A randomized, controlled trial. Montelukast/Beclomethasone Study Group. Ann Intern Med. 1999 Mar 16;130(6):487-95. doi: 10.7326/0003-4819-130-6-199903160-00005. PMID 10075616
- [Background] Damera G, Panettieri RA. Irreversible airway obstruction in asthma: what we lose, we lose early. Allergy Asthma Proc. 2014 Mar-Apr;35(2):111-8. doi: 10.2500/aap.2013.34.3724. PMID 24717787
- [Background] Bousquet J, Mantzouranis E, Cruz AA, Ait-Khaled N, Baena-Cagnani CE, Bleecker ER, Brightling CE, Burney P, Bush A, Busse WW, Casale TB, Chan-Yeung M, Chen R, Chowdhury B, Chung KF, Dahl R, Drazen JM, Fabbri LM, Holgate ST, Kauffmann F, Haahtela T, Khaltaev N, Kiley JP, Masjedi MR, Mohammad Y, O'Byrne P, Partridge MR, Rabe KF, Togias A, van Weel C, Wenzel S, Zhong N, Zuberbier T. Uniform definition of asthma severity, control, and exacerbations: document presented for the World Health Organization Consultation on Severe Asthma. J Allergy Clin Immunol. 2010 Nov;126(5):926-38. doi: 10.1016/j.jaci.2010.07.019. PMID 20926125
- [Background] Pelaia G, Vatrella A, Maselli R. The potential of biologics for the treatment of asthma. Nat Rev Drug Discov. 2012 Dec;11(12):958-72. doi: 10.1038/nrd3792. PMID 23197041
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Background] Jia G, Erickson RW, Choy DF, Mosesova S, Wu LC, Solberg OD, Shikotra A, Carter R, Audusseau S, Hamid Q, Bradding P, Fahy JV, Woodruff PG, Harris JM, Arron JR; Bronchoscopic Exploratory Research Study of Biomarkers in Corticosteroid-refractory Asthma (BOBCAT) Study Group. Periostin is a systemic biomarker of eosinophilic airway inflammation in asthmatic patients. J Allergy Clin Immunol. 2012 Sep;130(3):647-654.e10. doi: 10.1016/j.jaci.2012.06.025. Epub 2012 Aug 1. PMID 22857879
- [Background] Lai T, Wang S, Xu Z, Zhang C, Zhao Y, Hu Y, Cao C, Ying S, Chen Z, Li W, Wu B, Shen H. Long-term efficacy and safety of omalizumab in patients with persistent uncontrolled allergic asthma: a systematic review and meta-analysis. Sci Rep. 2015 Feb 3;5:8191. doi: 10.1038/srep08191. PMID 25645133
- [Background] Peirsman EJ, Carvelli TJ, Hage PY, Hanssens LS, Pattyn L, Raes MM, Sauer KA, Vermeulen F, Desager KN. Exhaled nitric oxide in childhood allergic asthma management: a randomised controlled trial. Pediatr Pulmonol. 2014 Jul;49(7):624-31. doi: 10.1002/ppul.22873. Epub 2013 Sep 4. PMID 24039119
- [Background] Anderson WJ, Short PM, Williamson PA, Lipworth BJ. Inhaled corticosteroid dose response using domiciliary exhaled nitric oxide in persistent asthma: the FENOtype trial. Chest. 2012 Dec;142(6):1553-1561. doi: 10.1378/chest.12-1310. PMID 23364390
- [Background] Gupta N, Su X, Popov B, Lee JW, Serikov V, Matthay MA. Intrapulmonary delivery of bone marrow-derived mesenchymal stem cells improves survival and attenuates endotoxin-induced acute lung injury in mice. J Immunol. 2007 Aug 1;179(3):1855-63. doi: 10.4049/jimmunol.179.3.1855. PMID 17641052
- [Background] Lee JW, Fang X, Gupta N, Serikov V, Matthay MA. Allogeneic human mesenchymal stem cells for treatment of E. coli endotoxin-induced acute lung injury in the ex vivo perfused human lung. Proc Natl Acad Sci U S A. 2009 Sep 22;106(38):16357-62. doi: 10.1073/pnas.0907996106. Epub 2009 Aug 31. PMID 19721001
- [Background] Fang X, Neyrinck AP, Matthay MA, Lee JW. Allogeneic human mesenchymal stem cells restore epithelial protein permeability in cultured human alveolar type II cells by secretion of angiopoietin-1. J Biol Chem. 2010 Aug 20;285(34):26211-22. doi: 10.1074/jbc.M110.119917. Epub 2010 Jun 16. PMID 20554518
- [Background] Gupta N, Krasnodembskaya A, Kapetanaki M, Mouded M, Tan X, Serikov V, Matthay MA. Mesenchymal stem cells enhance survival and bacterial clearance in murine Escherichia coli pneumonia. Thorax. 2012 Jun;67(6):533-9. doi: 10.1136/thoraxjnl-2011-201176. Epub 2012 Jan 16. PMID 22250097
- [Background] Krasnodembskaya A, Samarani G, Song Y, Zhuo H, Su X, Lee JW, Gupta N, Petrini M, Matthay MA. Human mesenchymal stem cells reduce mortality and bacteremia in gram-negative sepsis in mice in part by enhancing the phagocytic activity of blood monocytes. Am J Physiol Lung Cell Mol Physiol. 2012 May 15;302(10):L1003-13. doi: 10.1152/ajplung.00180.2011. Epub 2012 Mar 16. PMID 22427530
- [Background] Krasnodembskaya A, Song Y, Fang X, Gupta N, Serikov V, Lee JW, Matthay MA. Antibacterial effect of human mesenchymal stem cells is mediated in part from secretion of the antimicrobial peptide LL-37. Stem Cells. 2010 Dec;28(12):2229-38. doi: 10.1002/stem.544. PMID 20945332
- [Background] Lee JW, Krasnodembskaya A, McKenna DH, Song Y, Abbott J, Matthay MA. Therapeutic effects of human mesenchymal stem cells in ex vivo human lungs injured with live bacteria. Am J Respir Crit Care Med. 2013 Apr 1;187(7):751-60. doi: 10.1164/rccm.201206-0990OC. PMID 23292883
- [Background] Nemeth K, Leelahavanichkul A, Yuen PS, Mayer B, Parmelee A, Doi K, Robey PG, Leelahavanichkul K, Koller BH, Brown JM, Hu X, Jelinek I, Star RA, Mezey E. Bone marrow stromal cells attenuate sepsis via prostaglandin E(2)-dependent reprogramming of host macrophages to increase their interleukin-10 production. Nat Med. 2009 Jan;15(1):42-9. doi: 10.1038/nm.1905. Epub 2008 Nov 21. PMID 19098906
- [Background] Ortiz LA, Dutreil M, Fattman C, Pandey AC, Torres G, Go K, Phinney DG. Interleukin 1 receptor antagonist mediates the antiinflammatory and antifibrotic effect of mesenchymal stem cells during lung injury. Proc Natl Acad Sci U S A. 2007 Jun 26;104(26):11002-7. doi: 10.1073/pnas.0704421104. Epub 2007 Jun 14. PMID 17569781
- [Background] Mei SH, Haitsma JJ, Dos Santos CC, Deng Y, Lai PF, Slutsky AS, Liles WC, Stewart DJ. Mesenchymal stem cells reduce inflammation while enhancing bacterial clearance and improving survival in sepsis. Am J Respir Crit Care Med. 2010 Oct 15;182(8):1047-57. doi: 10.1164/rccm.201001-0010OC. Epub 2010 Jun 17. PMID 20558630
- [Background] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Background] Lee RH, Seo MJ, Reger RL, Spees JL, Pulin AA, Olson SD, Prockop DJ. Multipotent stromal cells from human marrow home to and promote repair of pancreatic islets and renal glomeruli in diabetic NOD/scid mice. Proc Natl Acad Sci U S A. 2006 Nov 14;103(46):17438-43. doi: 10.1073/pnas.0608249103. Epub 2006 Nov 6. PMID 17088535
- [Background] Parekkadan B, van Poll D, Suganuma K, Carter EA, Berthiaume F, Tilles AW, Yarmush ML. Mesenchymal stem cell-derived molecules reverse fulminant hepatic failure. PLoS One. 2007 Sep 26;2(9):e941. doi: 10.1371/journal.pone.0000941. PMID 17895982
- [Background] Togel F, Hu Z, Weiss K, Isaac J, Lange C, Westenfelder C. Administered mesenchymal stem cells protect against ischemic acute renal failure through differentiation-independent mechanisms. Am J Physiol Renal Physiol. 2005 Jul;289(1):F31-42. doi: 10.1152/ajprenal.00007.2005. Epub 2005 Feb 15. PMID 15713913
- [Background] Iso Y, Spees JL, Serrano C, Bakondi B, Pochampally R, Song YH, Sobel BE, Delafontaine P, Prockop DJ. Multipotent human stromal cells improve cardiac function after myocardial infarction in mice without long-term engraftment. Biochem Biophys Res Commun. 2007 Mar 16;354(3):700-6. doi: 10.1016/j.bbrc.2007.01.045. Epub 2007 Jan 17. PMID 17257581
- [Background] Schuleri KH, Feigenbaum GS, Centola M, Weiss ES, Zimmet JM, Turney J, Kellner J, Zviman MM, Hatzistergos KE, Detrick B, Conte JV, McNiece I, Steenbergen C, Lardo AC, Hare JM. Autologous mesenchymal stem cells produce reverse remodelling in chronic ischaemic cardiomyopathy. Eur Heart J. 2009 Nov;30(22):2722-32. doi: 10.1093/eurheartj/ehp265. Epub 2009 Jul 8. PMID 19586959
- [Background] Miyahara Y, Nagaya N, Kataoka M, Yanagawa B, Tanaka K, Hao H, Ishino K, Ishida H, Shimizu T, Kangawa K, Sano S, Okano T, Kitamura S, Mori H. Monolayered mesenchymal stem cells repair scarred myocardium after myocardial infarction. Nat Med. 2006 Apr;12(4):459-65. doi: 10.1038/nm1391. Epub 2006 Apr 2. PMID 16582917
- [Background] Hare JM, Traverse JH, Henry TD, Dib N, Strumpf RK, Schulman SP, Gerstenblith G, DeMaria AN, Denktas AE, Gammon RS, Hermiller JB Jr, Reisman MA, Schaer GL, Sherman W. A randomized, double-blind, placebo-controlled, dose-escalation study of intravenous adult human mesenchymal stem cells (prochymal) after acute myocardial infarction. J Am Coll Cardiol. 2009 Dec 8;54(24):2277-86. doi: 10.1016/j.jacc.2009.06.055. PMID 19958962
- [Background] Gong Z, Niklason LE. Use of human mesenchymal stem cells as alternative source of smooth muscle cells in vessel engineering. Methods Mol Biol. 2011;698:279-94. doi: 10.1007/978-1-60761-999-4_21. PMID 21431526
- [Background] Price AP, England KA, Matson AM, Blazar BR, Panoskaltsis-Mortari A. Development of a decellularized lung bioreactor system for bioengineering the lung: the matrix reloaded. Tissue Eng Part A. 2010 Aug;16(8):2581-91. doi: 10.1089/ten.TEA.2009.0659. PMID 20297903
- [Background] Deans RJ, Moseley AB. Mesenchymal stem cells: biology and potential clinical uses. Exp Hematol. 2000 Aug;28(8):875-84. doi: 10.1016/s0301-472x(00)00482-3. PMID 10989188
- [Background] Ishizawa K, Kubo H, Yamada M, Kobayashi S, Numasaki M, Ueda S, Suzuki T, Sasaki H. Bone marrow-derived cells contribute to lung regeneration after elastase-induced pulmonary emphysema. FEBS Lett. 2004 Jan 2;556(1-3):249-52. doi: 10.1016/s0014-5793(03)01399-1. PMID 14706858
- [Background] Spees JL, Pociask DA, Sullivan DE, Whitney MJ, Lasky JA, Prockop DJ, Brody AR. Engraftment of bone marrow progenitor cells in a rat model of asbestos-induced pulmonary fibrosis. Am J Respir Crit Care Med. 2007 Aug 15;176(4):385-94. doi: 10.1164/rccm.200607-1004OC. Epub 2007 May 11. PMID 17496228
- [Background] Spees JL, Whitney MJ, Sullivan DE, Lasky JA, Laboy M, Ylostalo J, Prockop DJ. Bone marrow progenitor cells contribute to repair and remodeling of the lung and heart in a rat model of progressive pulmonary hypertension. FASEB J. 2008 Apr;22(4):1226-36. doi: 10.1096/fj.07-8076com. Epub 2007 Nov 21. PMID 18032636
- [Background] Bonfield TL, Koloze M, Lennon DP, Zuchowski B, Yang SE, Caplan AI. Human mesenchymal stem cells suppress chronic airway inflammation in the murine ovalbumin asthma model. Am J Physiol Lung Cell Mol Physiol. 2010 Dec;299(6):L760-70. doi: 10.1152/ajplung.00182.2009. Epub 2010 Sep 3. PMID 20817776
- [Background] Lin HY, Xu L, Xie SS, Yu F, Hu HY, Song XL, Wang CH. Mesenchymal stem cells suppress lung inflammation and airway remodeling in chronic asthma rat model via PI3K/Akt signaling pathway. Int J Clin Exp Pathol. 2015 Aug 1;8(8):8958-67. eCollection 2015. PMID 26464637
- [Background] Trzil JE, Masseau I, Webb TL, Chang CH, Dodam JR, Liu H, Quimby JM, Dow SW, Reinero CR. Intravenous adipose-derived mesenchymal stem cell therapy for the treatment of feline asthma: a pilot study. J Feline Med Surg. 2016 Dec;18(12):981-990. doi: 10.1177/1098612X15604351. Epub 2015 Sep 17. PMID 26384398
- [Background] Gao J, Dennis JE, Muzic RF, Lundberg M, Caplan AI. The dynamic in vivo distribution of bone marrow-derived mesenchymal stem cells after infusion. Cells Tissues Organs. 2001;169(1):12-20. doi: 10.1159/000047856. PMID 11340257
- [Background] Cargnoni A, Gibelli L, Tosini A, Signoroni PB, Nassuato C, Arienti D, Lombardi G, Albertini A, Wengler GS, Parolini O. Transplantation of allogeneic and xenogeneic placenta-derived cells reduces bleomycin-induced lung fibrosis. Cell Transplant. 2009;18(4):405-22. doi: 10.3727/096368909788809857. PMID 19622228
- [Background] Moodley Y, Atienza D, Manuelpillai U, Samuel CS, Tchongue J, Ilancheran S, Boyd R, Trounson A. Human umbilical cord mesenchymal stem cells reduce fibrosis of bleomycin-induced lung injury. Am J Pathol. 2009 Jul;175(1):303-13. doi: 10.2353/ajpath.2009.080629. Epub 2009 Jun 4. PMID 19497992
- [Background] Lee SH, Jang AS, Kim YE, Cha JY, Kim TH, Jung S, Park SK, Lee YK, Won JH, Kim YH, Park CS. Modulation of cytokine and nitric oxide by mesenchymal stem cell transfer in lung injury/fibrosis. Respir Res. 2010 Feb 8;11(1):16. doi: 10.1186/1465-9921-11-16. PMID 20137099
- [Background] Rojas M, Xu J, Woods CR, Mora AL, Spears W, Roman J, Brigham KL. Bone marrow-derived mesenchymal stem cells in repair of the injured lung. Am J Respir Cell Mol Biol. 2005 Aug;33(2):145-52. doi: 10.1165/rcmb.2004-0330OC. Epub 2005 May 12. PMID 15891110
- [Background] Ortiz LA, Gambelli F, McBride C, Gaupp D, Baddoo M, Kaminski N, Phinney DG. Mesenchymal stem cell engraftment in lung is enhanced in response to bleomycin exposure and ameliorates its fibrotic effects. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8407-11. doi: 10.1073/pnas.1432929100. Epub 2003 Jun 18. PMID 12815096
- [Background] Jiang Y, Jahagirdar BN, Reinhardt RL, Schwartz RE, Keene CD, Ortiz-Gonzalez XR, Reyes M, Lenvik T, Lund T, Blackstad M, Du J, Aldrich S, Lisberg A, Low WC, Largaespada DA, Verfaillie CM. Pluripotency of mesenchymal stem cells derived from adult marrow. Nature. 2002 Jul 4;418(6893):41-9. doi: 10.1038/nature00870. Epub 2002 Jun 20. PMID 12077603
- [Background] Kotton DN, Ma BY, Cardoso WV, Sanderson EA, Summer RS, Williams MC, Fine A. Bone marrow-derived cells as progenitors of lung alveolar epithelium. Development. 2001 Dec;128(24):5181-8. doi: 10.1242/dev.128.24.5181. PMID 11748153
- [Background] Sueblinvong V, Loi R, Eisenhauer PL, Bernstein IM, Suratt BT, Spees JL, Weiss DJ. Derivation of lung epithelium from human cord blood-derived mesenchymal stem cells. Am J Respir Crit Care Med. 2008 Apr 1;177(7):701-11. doi: 10.1164/rccm.200706-859OC. Epub 2007 Dec 6. PMID 18063840
- [Background] Ma N, Gai H, Mei J, Ding FB, Bao CR, Nguyen DM, Zhong H. Bone marrow mesenchymal stem cells can differentiate into type II alveolar epithelial cells in vitro. Cell Biol Int. 2011 Dec;35(12):1261-6. doi: 10.1042/CBI20110026. PMID 21542803
- [Background] Yamada M, Kubo H, Kobayashi S, Ishizawa K, Numasaki M, Ueda S, Suzuki T, Sasaki H. Bone marrow-derived progenitor cells are important for lung repair after lipopolysaccharide-induced lung injury. J Immunol. 2004 Jan 15;172(2):1266-72. doi: 10.4049/jimmunol.172.2.1266. PMID 14707105
- [Background] Chang JC, Summer R, Sun X, Fitzsimmons K, Fine A. Evidence that bone marrow cells do not contribute to the alveolar epithelium. Am J Respir Cell Mol Biol. 2005 Oct;33(4):335-42. doi: 10.1165/rcmb.2005-0129OC. Epub 2005 Jun 16. PMID 15961725
- [Background] Kotton DN, Fabian AJ, Mulligan RC. Failure of bone marrow to reconstitute lung epithelium. Am J Respir Cell Mol Biol. 2005 Oct;33(4):328-34. doi: 10.1165/rcmb.2005-0175RC. Epub 2005 Jun 16. PMID 15961722
- [Background] Kumamoto M, Nishiwaki T, Matsuo N, Kimura H, Matsushima K. Minimally cultured bone marrow mesenchymal stem cells ameliorate fibrotic lung injury. Eur Respir J. 2009 Sep;34(3):740-8. doi: 10.1183/09031936.00128508. Epub 2009 Mar 26. PMID 19324956
- [Background] Bitencourt CS, Pereira PA, Ramos SG, Sampaio SV, Arantes EC, Aronoff DM, Faccioli LH. Hyaluronidase recruits mesenchymal-like cells to the lung and ameliorates fibrosis. Fibrogenesis Tissue Repair. 2011 Jan 13;4(1):3. doi: 10.1186/1755-1536-4-3. PMID 21232095
- [Background] Tashiro J, Elliot SJ, Gerth DJ, Xia X, Pereira-Simon S, Choi R, Catanuto P, Shahzeidi S, Toonkel RL, Shah RH, El Salem F, Glassberg MK. Therapeutic benefits of young, but not old, adipose-derived mesenchymal stem cells in a chronic mouse model of bleomycin-induced pulmonary fibrosis. Transl Res. 2015 Dec;166(6):554-67. doi: 10.1016/j.trsl.2015.09.004. Epub 2015 Sep 18. PMID 26432923
- [Background] Lee SH, Lee EJ, Lee SY, Kim JH, Shim JJ, Shin C, In KH, Kang KH, Uhm CS, Kim HK, Yang KS, Park S, Kim HS, Kim YM, Yoo TJ. The effect of adipose stem cell therapy on pulmonary fibrosis induced by repetitive intratracheal bleomycin in mice. Exp Lung Res. 2014 Apr;40(3):117-25. doi: 10.3109/01902148.2014.881930. PMID 24624895
- [Background] Royce SG, Shen M, Patel KP, Huuskes BM, Ricardo SD, Samuel CS. Mesenchymal stem cells and serelaxin synergistically abrogate established airway fibrosis in an experimental model of chronic allergic airways disease. Stem Cell Res. 2015 Nov;15(3):495-505. doi: 10.1016/j.scr.2015.09.007. Epub 2015 Sep 25. PMID 26426509
- [Background] Xu J, Mora A, Shim H, Stecenko A, Brigham KL, Rojas M. Role of the SDF-1/CXCR4 axis in the pathogenesis of lung injury and fibrosis. Am J Respir Cell Mol Biol. 2007 Sep;37(3):291-9. doi: 10.1165/rcmb.2006-0187OC. Epub 2007 Apr 26. PMID 17463394
- [Background] Antoniou KM, Papadaki HA, Soufla G, Kastrinaki MC, Damianaki A, Koutala H, Spandidos DA, Siafakas NM. Investigation of bone marrow mesenchymal stem cells (BM MSCs) involvement in Idiopathic Pulmonary Fibrosis (IPF). Respir Med. 2010 Oct;104(10):1535-42. doi: 10.1016/j.rmed.2010.04.015. Epub 2010 May 18. PMID 20483575
- [Background] Wilson JG, Liu KD, Zhuo H, Caballero L, McMillan M, Fang X, Cosgrove K, Vojnik R, Calfee CS, Lee JW, Rogers AJ, Levitt J, Wiener-Kronish J, Bajwa EK, Leavitt A, McKenna D, Thompson BT, Matthay MA. Mesenchymal stem (stromal) cells for treatment of ARDS: a phase 1 clinical trial. Lancet Respir Med. 2015 Jan;3(1):24-32. doi: 10.1016/S2213-2600(14)70291-7. Epub 2014 Dec 17. PMID 25529339
- [Background] Liang J, Zhang H, Hua B, Wang H, Lu L, Shi S, Hou Y, Zeng X, Gilkeson GS, Sun L. Allogenic mesenchymal stem cells transplantation in refractory systemic lupus erythematosus: a pilot clinical study. Ann Rheum Dis. 2010 Aug;69(8):1423-9. doi: 10.1136/ard.2009.123463. PMID 20650877
- [Background] Weiss DJ, Casaburi R, Flannery R, LeRoux-Williams M, Tashkin DP. A placebo-controlled, randomized trial of mesenchymal stem cells in COPD. Chest. 2013 Jun;143(6):1590-1598. doi: 10.1378/chest.12-2094. PMID 23172272
- [Background] Chambers DC, Enever D, Ilic N, Sparks L, Whitelaw K, Ayres J, Yerkovich ST, Khalil D, Atkinson KM, Hopkins PM. A phase 1b study of placenta-derived mesenchymal stromal cells in patients with idiopathic pulmonary fibrosis. Respirology. 2014 Oct;19(7):1013-8. doi: 10.1111/resp.12343. Epub 2014 Jul 9. PMID 25039426
- [Background] Tzouvelekis A, Paspaliaris V, Koliakos G, Ntolios P, Bouros E, Oikonomou A, Zissimopoulos A, Boussios N, Dardzinski B, Gritzalis D, Antoniadis A, Froudarakis M, Kolios G, Bouros D. A prospective, non-randomized, no placebo-controlled, phase Ib clinical trial to study the safety of the adipose derived stromal cells-stromal vascular fraction in idiopathic pulmonary fibrosis. J Transl Med. 2013 Jul 15;11:171. doi: 10.1186/1479-5876-11-171. PMID 23855653
- [Background] Weiss DJ, Chambers D, Giangreco A, Keating A, Kotton D, Lelkes PI, Wagner DE, Prockop DJ; ATS Subcommittee on Stem Cells and Cell Therapies. An official American Thoracic Society workshop report: stem cells and cell therapies in lung biology and diseases. Ann Am Thorac Soc. 2015 Apr;12(4):S79-97. doi: 10.1513/AnnalsATS.201502-086ST. PMID 25897748
- [Background] Glassberg MK, Toonkel RL. Moving stem cell therapy to patients with idiopathic pulmonary fibrosis. Respirology. 2014 Oct;19(7):950-1. doi: 10.1111/resp.12364. Epub 2014 Aug 14. No abstract available. PMID 25124287
- [Background] Toonkel RL, Hare JM, Matthay MA, Glassberg MK. Mesenchymal stem cells and idiopathic pulmonary fibrosis. Potential for clinical testing. Am J Respir Crit Care Med. 2013 Jul 15;188(2):133-40. doi: 10.1164/rccm.201207-1204PP. PMID 23306542
- [Background] Hare JM, Fishman JE, Gerstenblith G, DiFede Velazquez DL, Zambrano JP, Suncion VY, Tracy M, Ghersin E, Johnston PV, Brinker JA, Breton E, Davis-Sproul J, Schulman IH, Byrnes J, Mendizabal AM, Lowery MH, Rouy D, Altman P, Wong Po Foo C, Ruiz P, Amador A, Da Silva J, McNiece IK, Heldman AW, George R, Lardo A. Comparison of allogeneic vs autologous bone marrow-derived mesenchymal stem cells delivered by transendocardial injection in patients with ischemic cardiomyopathy: the POSEIDON randomized trial. JAMA. 2012 Dec 12;308(22):2369-79. doi: 10.1001/jama.2012.25321. PMID 23117550
- [Background] Sundin M, Orvell C, Rasmusson I, Sundberg B, Ringden O, Le Blanc K. Mesenchymal stem cells are susceptible to human herpesviruses, but viral DNA cannot be detected in the healthy seropositive individual. Bone Marrow Transplant. 2006 Jun;37(11):1051-9. doi: 10.1038/sj.bmt.1705368. PMID 16604097
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Jia CE, Zhang HP, Lv Y, Liang R, Jiang YQ, Powell H, Fu JJ, Wang L, Gibson PG, Wang G. The Asthma Control Test and Asthma Control Questionnaire for assessing asthma control: Systematic review and meta-analysis. J Allergy Clin Immunol. 2013 Mar;131(3):695-703. doi: 10.1016/j.jaci.2012.08.023. Epub 2012 Oct 8. PMID 23058645
- [Background] Klyushnenkova E, Mosca JD, Zernetkina V, Majumdar MK, Beggs KJ, Simonetti DW, Deans RJ, McIntosh KR. T cell responses to allogeneic human mesenchymal stem cells: immunogenicity, tolerance, and suppression. J Biomed Sci. 2005;12(1):47-57. doi: 10.1007/s11373-004-8183-7. PMID 15864738
- [Background] Le Blanc K, Tammik C, Rosendahl K, Zetterberg E, Ringden O. HLA expression and immunologic properties of differentiated and undifferentiated mesenchymal stem cells. Exp Hematol. 2003 Oct;31(10):890-6. doi: 10.1016/s0301-472x(03)00110-3. PMID 14550804
- See also: Global Initiative for Asthma 2015 from the Global Strategy for Asthma Management and Prevention — http://www.ginasthma.org